CLINICAL TRIAL: NCT01897259
Title: Comparison of Conservative Methods for the Treatment of Lateral Epicondylitis: A Randomized, Prospective Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11.0566
Record Dates: First submitted 2012-06-11; First posted 2013-07-11 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
Keywords: tennis elbow; lateral epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Physical Therapy Modalities; Prolotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Corticosteroid Injections (Active Comparator): Patients will receive 1 cc Kenalong 10 mg injection to the site every 6 weeks until clinical symptoms have resolved. They will also receive an anesthetic of 1cc 1% lidocaine in conjunction with the corticosteroid injection.
  Interventions: Drug: Corticosteroid Injections
- Prolotherapy (Active Comparator): Participants receive 1cc 50% Dextrose and 1 cc Sodium Morrhuate to the site every 6 weeks until symptoms resolve. These participants will also receive an anesthetic of 1cc 1% lidocaine.
  Interventions: Drug: Prolotherapy
- Placebo (Placebo Comparator): Participants will recieve placebo injections (1cc 1% lidocaine and 1cc normal saline).
  Interventions: Drug: Placebo Injection
- Physical Therapy (Active Comparator): Participants will be prescribed NSAIDS (Diclofenac 75 mg BID) for 2 weeks. Participants will attend therapy for muscle stretches, soft tissue mobilization, and gradual strengthening.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Drug: Placebo Injection — Participants in the placebo group will recieve placebo injections (1cc 1% lidocaine and 1cc normal saline).
  Arms: Placebo
Behavioral: Physical Therapy — Subjects participating in the physical therapy group will attend physical therapy and be prescribed to NSAIDS. No prolotherapy or corticosteroid injections.
  Arms: Physical Therapy
Drug: Corticosteroid Injections — Participants in the corticosteroid group will recieve corticosteroid injections (1 cc Kenalog 10 mg). They will also recieve anesthetic of 1 ml 1% lidocaine.
  Arms: Corticosteroid Injections
Drug: Prolotherapy — Subjects participating in the prolotherapy group will recieve 1 cc 50% Dextrose and Sodium Morrhuate 1 cc injections.
  Arms: Prolotherapy

SUMMARY:
This is a prospective study where patients with lateral epicondylitis (tennis elbow) will be randomized into one of 4 possible treatments. The purpose is to individually examine the efficacy of each treatment, and determine if one treatment method is more effective than another. The four treatments are: corticosteriod injections, prolotherapy, NSAIDs (non-steroidal anti-inflammatory drugs) combined with physical therapy, and a placebo.

ELIGIBILITY:
Inclusion Criteria:

* pain over the lateral epicondyle (via palpation over the lateral epicondyle, resisted wrist extension, resisted finger extension of the middle finger) for less than six-months duration prior to enrollment
* conservative treatment of tennis elbow is recommended as standard of care treatment
* over the age of 18 and under the age of 65
* ability to give informed consent

Exclusion Criteria:

* treatment by a health care profession (MD, physicians assistnat, therapist, or nurse practitioner) within the previous 6 months for tennis elbow
* congenital deformities, tendon ruptures, or fractures of the elbow within the previous 12 months
* immobility casts or splints within the last 6 months for tennis elbow
* co-existing elbow diagnosis (i.e. osteoarthritis or instability)
* pregnant women, women trying to get pregnant, or breastfeeding women
* under the age of 18 or over the age of 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Symptom Severity in pre intervention assessments | 12 months
Symptom severity in post-intervention assessments | 12 months

SECONDARY OUTCOMES:
Functional status score pre-intervention | 12 months
  The secondary outcome will be by means of functional status score by means of QuickDASH (Disabilities of Arm, Shoulder, and Hand) prior to intervention.
Functional status score severity- post intervention | 12 months
  The secondary outcome will be the functional status score by means of the QuickDash (Disabilities of Arm, Shoulder and Hand) for post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tuna Ozyurekoglu, MD, Principal Investigator — Christine M. Kleinert Institute for Hand and Microsurgery
Locations (1):
- Christine M. Kleinert Institute of Hand and Microsurgery, Louisville, Kentucky, United States